CLINICAL TRIAL: NCT01204203
Title: A Pilot Phase 2 Study of Bisphosphonate Therapy (Zoledronic Acid) in Patients With Advanced Malignant Mesothelioma
Brief Title: Pilot Study of Bisphosphonate Therapy (Zoledronic Acid) in Patients With Malignant Mesothelioma (UAB 0901)
Acronym: UAB0901
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Francisco Robert,MD, Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F090917002 (UAB 0901); UAB 0901 (Other Grant/Funding Number: Novartis CZOL446EUS144T)
Record Dates: First submitted 2010-09-15; First posted 2010-09-17 (Estimated); Results first posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-04

CONDITIONS: Mesothelioma
Keywords: mesothelioma; zoledronic acid; zometa; bisphosphonate therapy; CT scan; PET scan
MeSH Terms: conditions — Mesothelioma | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Zometa (Experimental): Zometa (zoledronic acid) will be administered by infusion on Day 1 of a 3-week cycle followed by tumor assessment from CT and/or PET scans every 2 cycles. This will continue until progression of disease and/or intolerable toxicity.
  Interventions: Drug: Zometa

INTERVENTIONS:
Drug: Zometa — Zoledronic acid will be administered IV on the first day of a 21 day cycle at a concentration of 4 mg. The treatment will take about 30-60 minutes with the infusion lasting about 15 minutes.
  Other Names: Zoledronic acid

SUMMARY:
The primary objective of this trial is to determine the response rate of single agent zoledronic acid using a composite of criteria including the EORTC modified RECIST criteria and the EORTC tumor response criteria for 18F-FDG PET scans.

DETAILED DESCRIPTION:
This pilot study will examine the effect of bisphosphonate (zoledronic acid) in patients with malignant mesothelioma. Evaluation will be limited to patients with standard (CT scans) and functional instruments (FDG PET Scans) of tumor assessment after the administration of standard doses of zoledronic acid (4 mg IV every 3 weeks). We will also explore the biologic effect of zoledronic acid in patients using new serum markers as well as several blood level markers.

ELIGIBILITY:
Inclusion Criteria:

* Males and females > 18 years of age
* Life expectancy of at least 2 months
* Histologically confirmed unresectable malignant pleural mesothelioma (MPM)
* Measurable disease by CT Scan criteria and/or positive metabolic activity of 18F-FDG PET Scan criteria at screening
* ECOG Performance Status of 0-2
* Laboratory and clinical results within 2 weeks prior to Day 1 must be as follows:

  1. ANC ≥ 1.5 x 109/L
  2. Platelet Count ≥ 100 x 109/L
  3. Hemoglobin ≥ 9g/dL
  4. Serum bilirubin ≤ 1.5 x upper limit of normal (ULN)
  5. AST ≤ 2.5 x ULN
  6. ALT ≤ 2.5 x ULN
  7. ALK-P ≤ 3 x ULN
  8. Serum creatinine ≤ 1.8mg/dL
  9. Calculated Serum Creatinine Clearance 40 - > 60ml/min
* Female subjects of childbearing potential and all male subjects must be surgically sterile or consent to use a medically acceptable method of contraception throughout the trial.
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Known central nervous system (CNS) tumor involvement
* Evidence of other active malignancy requiring treatment
* Clinically significant heart disease (e.g., congestive heart failure of New York Heart Association Class 3 or 4 angina not well controlled by medication, or myocardial infarction within 6 months)
* Known infection with HIV or hepatitis
* Clinically significant arrhythmias demonstrated on electrocardiogram (ECG). Note: subjects with chronic atrial arrhythmia, i.e., atrial fibrillation or paroxysmal supraventricular tachycardia (SVT) are eligible.
* Active, serious systemic disease, including active bacterial or fungal infection.
* Subjects undergoing invasive dental procedures, significant periodontal disease or history of osteonecrosis of the jaw.
* Treatment within 4 weeks of the start of the trial with other systemic anticancer therapy.
* Breastfeeding, pregnant, or likely to become pregnant during the clinical trial.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-06; Primary Completion 2015-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Robert, M.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Inclusion criteria included: adult patients (age>18) with unresectable Malignant Pleural Mesothelioma (MPM) who had progressed after one or more prior systemic therapies, had not received prior systemic therapy due to poor performance status (PS), and/or were unwilling to receive systemic chemotherapy.
Pre-assignment Details: The primary objective of this study was to evaluate the anti-tumor activity of zoledronic acid (Zometa) in subjects with unresectable, advanced Malignant Pleural Mesothelioma (MPM).
Groups:
- Zoledronic Acid (Zometa): Zoledronic acid (Zometa) will be administered by infusion on Day 1 of a 3-week cycle followed by tumor assessment from CT and/or PET scans every 2 cycles. This will continue until progression of disease and/or intolerable toxicity.
  Zoledronic acid (Zometa) will be administered IV on the first day of a 21 day cycle at a concentration of 4 mg. The treatment will take about 30-60 minutes with the infusion lasting about 15 minutes.
Period: Overall Study
Arm/Group | Zoledronic Acid (Zometa)
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Zoledronic Acid (Zometa): Zometa (zoledronic acid) 4mg will be administered by infusion on Day 1 of a 3-week cycle followed by tumor assessment from CT and/or PET scans every 2 cycles. This will continue until progression of disease and/or intolerable toxicity.
Arm/Group | Zoledronic Acid (Zometa)
Number analyzed (Participants) | 8
Age, Continuous [Median (Full Range); unit: years] | 62 [49 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response Rate Following Zoledronic Acid (Zometa)
Description: The modified Response Evaluation Criteria in Solid Tumors Criteria (RECIST 2004) will be used for target lesions and assessed by CT scans. Complete Response (CR) is the disappearance of target lesions; Partial Response (PR) is greater than or equal to 30% reduction in the total tumor measurement; Stable Disease (SD) is the absence of response or progression; and Progressive Disease (PD) is a 20% increase in the total tumor measurement over nadir value or the appearance of new lesions.
Time Frame: Baseline up to 28 months or until progressive disease or death
Population: Participants with advanced malignant pleural mesothelioma.
Measure: Number; unit: percentage of responders
Arm/Group | Zometa
Number analyzed (Participants) | 8
percentage of responders | 12.5

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression Free Survival is defined as the number of days from the day the subject started treatment to the day the subject experienced evidence of disease progression, as determined by radiological or clinical progression.
Time Frame: Baseline up to 28 months
Population: Participants with advanced malignant pleural mesothelioma.
Measure: Median (Full Range); unit: Months
Arm/Group | Zometa
Number analyzed (Participants) | 8
Months | 2 [0.5 to 21]

3. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival is defined as the number of days from the day the subject started treatment to the day the subject experienced death or lost to follow-up.
Time Frame: Baseline up to 28 months
Population: Participants with advanced malignant pleural mesothelioma.
Measure: Median (Full Range); unit: months
Arm/Group | Zometa
Number analyzed (Participants) | 8
months | 7 [0.8 to 28]

ADVERSE EVENTS:
Time Frame: From baseline to 28 months
Description: Subjects with either stable disease or objective response continued treatment until disease progression and/or intolerable toxicity at which patients were taken off study. Subjects were monitored for toxicity using NCI CTAE v3.0 Criteria. Dose adjustment was allowed per standard guidelines for zoledronic acid for decreased creatinine clearance. Patients who completed at least one treatment cycle were included in data analysis.
Groups:
- Zoledronic Acid (Zometa): Zoledronic acid (Zometa) will be administered IV-4mg by infusion on Day 1 of a 3-week cycle followed by tumor assessment from CT and/or PET scans every 2 cycles.The treatment will take about 30-60 minutes with the infusion lasting about 15 minutes.This will continue until progression of disease and/or intolerable toxicity.
Arm/Group | Zoledronic Acid (Zometa)
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No